CLINICAL TRIAL: NCT04140734
Title: Study Protocol for Comparison of Lower Eyelid Retraction Repair With Hard Palate, Autologous Ear Cartilage, and Porcine Acellular Dermal Matrix Spacer Grafts
Brief Title: Spacer Graft Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-10410
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Eyelid Diseases; Eyelid Droop
Keywords: Retraction Repair; Hard Palate; Autologous Ear Cartilage; porcine acellular dermal matrix; spacer graft
MeSH Terms: conditions — Eyelid Diseases; Blepharoptosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Hard Palate (Experimental): Some patients who will already be undergoing lower eyelid retraction repair with a spacer graft will be randomized to use hard palate
  Interventions: Device: Spacer Graft
- Autologous Ear Cartilage (Experimental): Some patients who will already be undergoing lower eyelid retraction repair with a spacer graft will be randomized to use autologous ear cartilage
  Interventions: Device: Spacer Graft
- Porcine Acellular Dermal Matrix (Experimental): Some patients who will already be undergoing lower eyelid retraction repair with a spacer graft will be randomized to use porcine acellular dermal matrix
  Interventions: Device: Spacer Graft

INTERVENTIONS:
Device: Spacer Graft — In this prospective, randomized clinical trial, patients who will already be undergoing lower eyelid retraction repair with a spacer graft will randomly be assigned via a randomization web-site to receive 1 of 3 spacer grafts: hard palate, autologous auricular cartilage, and porcine acellular dermal matrix (Enduragen). Both the patient and the surgeon will know which of the three possible grafts are being used.

SUMMARY:
To determine which of three types of spacer grafts (hard palate vs autologous ear cartilage vs Enduragen) are the most effective in lower eyelid retraction repair outcomes as measured by MRD2 (margin to reflex distance 2)

DETAILED DESCRIPTION:
Lower eyelid retraction is a common eyelid malposition, typically caused by thyroid eye disease, excessive resection of skin in a cosmetic lower eyelid blepharoplasty, vertical rectus muscle recession, facial nerve paralysis, or a normal anatomical variant. When the lower eyelid is displaced inferiorly, exposing sclera between the limbus and the eyelid margin, symptoms can vary from ocular irritation and discomfort to vision threatening corneal decompensation. If medical management does not suffice, surgery is indicated.

Although lower eyelid retractor lysis alone has been described, supporting material (spacer graft) placed to augment the posterior lamella is generally required for more effective elevation of the eyelid. Various materials have been utilized, including autologous auricular cartilage, bovine acellular dermal matrix, porcine acellular dermal matrix, hard palate mucosa, dermis and dermis fat grafts. Previous studies on acellular dermal matrix use in lower eyelid retraction repair consist of retrospective efficacy studies with only 2 comparative studies. However, conflicting results raised doubt as to which material was superior. In addition, a prospective, randomized comparative study of spacer grafts used for lower eyelid retraction repair was done comparing autologous auricular cartilage, porcine acellular dermal matrix, and bovine acellular dermal matrix. The results yielded no statistically significant difference in surgical outcomes and complications. As of now, surgery with any of the spacer grafts, including autologous hard palate, is accepted as standard of care.

This study is designed to determine whether using hard palate as a spacer graft will have statistically significant different surgical outcomes and complications as compared to autologous ear cartilage and porcine acellular dermal matrix spacer grafts. Although studied separately, this has not been studied before in a prospective randomized manner and may prove to demonstrate improved surgical results and decreased complications. This can guide future choice of spacer graft used in lower eyelid retraction repair surgery.

ELIGIBILITY:
Inclusion Criteria:

* Underwent lower eyelid retraction repair requiring a spacer graft between July 1, 2019 and July 1, 2022

Exclusion Criteria:

* Younger than 18 years old
* Required concurrent surgeries (e.g., midface lift or full thickness skin graft) or required further surgeries on the operated eyelid within the 6 months postoperatively
* Patients with less than 1-month follow up will be excluded from all outcome analysis and those without postoperative 6-month data will be excluded from the postoperative month 6 MRD2 calculation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Lower Eyelid Height | Preoperatively, and at 1 week, 1 month, 3 months and 6 months post-operatively
  Lower Eyelid Height will be measured via Margin Reflect Distance 2 (MRD2). Photographs taken during study visits will analyze the effectiveness of the spacer grafts with respect to lower eyelid retraction repair. MRD2 is the distance in millimeters between the pupillary light reflex and the lower eyelid margin with the patient looking at a light reflex in primary gaze. Results will be summarized and reported by study arm using basic descriptive statistics. A normal MRD2 is about 4. The higher the number for MRD2, the more severe the retraction. Postoperatively, a lower MRD2 indicates a better surgical outcome.

SECONDARY OUTCOMES:
Post-Surgical Complications | Preoperatively, and at 1 week, 1 month, 3 months and 6 months post-operatively
  Post-Surgical Complications will be summarized using specific complications as graded by either the examiner or the patient. Specifically, conjunctival injection and eyelid swelling will be graded by the examiner on a scale of 0 to 10 where "0" indicates no visible injection or swelling (normal), respectively and "10" is indicative of the most severe level of conjuctival redness or swelling, respectively. Similarly, tearing, itching, and discomfort will be individually graded by the patient on a scale of 0-10 wherein "0" is indicative of no tearing, itching, or discomfort, respectively and "10" is indicative of maximal tearing, itching, and discomfort, respectively. Results will be summarized and reported by study arm using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Barmettler, MD, Principal Investigator — Director of Oculoplastic Surgery Division
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartley GB. The differential diagnosis and classification of eyelid retraction. Ophthalmology. 1996 Jan;103(1):168-76. doi: 10.1016/s0161-6420(96)30744-6. PMID 8628549
- [Background] Baylis HI, Nelson ER, Goldberg RA. Lower eyelid retraction following blepharoplasty. Ophthalmic Plast Reconstr Surg. 1992;8(3):170-5. doi: 10.1097/00002341-199209000-00002. PMID 1390423
- [Background] Barmettler A, Heo M. A Prospective, Randomized Comparison of Lower Eyelid Retraction Repair With Autologous Auricular Cartilage, Bovine Acellular Dermal Matrix (Surgimend), and Porcine Acellular Dermal Matrix (Enduragen) Spacer Grafts. Ophthalmic Plast Reconstr Surg. 2018 May/Jun;34(3):266-273. doi: 10.1097/IOP.0000000000000946. PMID 28658181
- [Background] Wearne MJ, Sandy C, Rose GE, Pitts J, Collin JR. Autogenous hard palate mucosa: the ideal lower eyelid spacer? Br J Ophthalmol. 2001 Oct;85(10):1183-7. doi: 10.1136/bjo.85.10.1183. PMID 11567962
- [Background] Liao YL, Wu SY, Tsai YJ. Long-Term Results of Autologous Auricular Cartilage Graft Applied in Anophthalmic Orbits Unable to Wear Prosthesis. J Ophthalmol. 2019 Apr 9;2019:7197063. doi: 10.1155/2019/7197063. eCollection 2019. PMID 31093371